CLINICAL TRIAL: NCT01861262
Title: Percentage of Oxygen Saturation of Haemoglobin in Tissues (StO2) Performance Measured on Admission to the Emergency Department in the Assessment of Drug Poisoning
Brief Title: StO2 Performance Measured on Admission to the Emergency Department in the Assessment of Drug Poisoning
Acronym: IMACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12 506 03
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Drug Poisoning
Keywords: emergency; drug poisoning; StO2 measurement; blood pressure; hemodynamic failure
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Measurement of StO2 (Experimental): The procedure is a measurement and non-invasive monitoring system of percentage of oxygen saturation of haemoglobin in tissues using infrared technology. The system used in the study is the tissue oxygenation monitor InSpectraTM StO2 Spot Check, Model 300 consisting of a clamp applied to the base of the thumb of the patient.
  Interventions: Device: Measurement of StO2

INTERVENTIONS:
Device: Measurement of StO2 — The procedure is a measurement and non-invasive monitoring system of percentage of oxygen saturation of haemoglobin in tissues using infrared technology. The system used in the study is the tissue oxygenation monitor InSpectraTM StO2 Spot Check, Model 300 consisting of a clamp applied to the base of the thumb of the patient.

SUMMARY:
The primary purpose of the protocol is to evaluate the StO2 performance measured at the admission to the emergency department to identify hemodynamic failure at the admission or within the first three hours of monitoring patients with drug poisoning.

The study hypotheses are:

* The early detection of hypoperfusion by StO2, essential to prevent the development of collapse.
* To limit hemodynamic failure effects, reduce morbidity and mortality of drug poisoning, hospital stay and cost.

DETAILED DESCRIPTION:
The procedure is a measurement and non-invasive monitoring system of percentage of oxygen saturation of haemoglobin in tissues using infrared technology. The system used in the study is the tissue oxygenation monitor InSpectraTM StO2 Spot Check, Model 300 consisting of a clamp applied to the base of the thumb of the patient.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the emergency department,
* whose pattern of hospitalization is drug poisoning, defined on data from the patient's interrogation or his family if the patient is not able to answer,
* Written informed consent signed by the patient or, if he's unable to sign, by a companion,
* Affiliated to medical insurance

Exclusion Criteria:

* Patients without thenar eminence or having a disease of the thenar,
* Refusal to participate in the study,
* Participation in another biomedical research,
* Patient under guardianship, trusteeship or judicial protection,
* Pregnant women or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
StO2 performance measured to identify hemodynamic failure. | Outcome measure is assessed during three hours after the admission to the emergency department.

SECONDARY OUTCOMES:
StO2 distribution | Outcome measure is assessed during three hours after the admission to the emergency department.
StO2 threshold value to predict the onset of hemodynamic failure | Outcome measure is assessed during three hours after the admission to the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie DEHOURS, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, Midi-Pyrenees, France

REFERENCES:
- [Background] Lambert H, Manel J, Bellou A, el Kouch S. [Morbidity and mortality from acute drug poisoning in France]. Rev Prat. 1997 Apr 1;47(7):716-20. French. PMID 9183946
- [Background] F.Adnet, S.Atout, M. Galinski. Evolution des intoxications médicamenteuses volontaires en France, 2005, Société de réanimation de langue française
- [Background] Cohn SM, Nathens AB, Moore FA, Rhee P, Puyana JC, Moore EE, Beilman GJ; StO2 in Trauma Patients Trial Investigators. Tissue oxygen saturation predicts the development of organ dysfunction during traumatic shock resuscitation. J Trauma. 2007 Jan;62(1):44-54; discussion 54-5. doi: 10.1097/TA.0b013e31802eb817. PMID 17215732
- [Background] Reducing the severity of road injuries through post impact care. European Transport Safety Council. Eur J Emerg Med. 1999 Sep;6(3):271-4. doi: 10.1097/00063110-199909000-00020. No abstract available. PMID 10622398
- [Background] Cohn SM, Crookes BA, Proctor KG. Near-infrared spectroscopy in resuscitation. J Trauma. 2003 May;54(5 Suppl):S199-202. doi: 10.1097/01.TA.0000047225.53051.7C. No abstract available. PMID 12768125
- [Background] Crookes BA, Cohn SM, Bloch S, Amortegui J, Manning R, Li P, Proctor MS, Hallal A, Blackbourne LH, Benjamin R, Soffer D, Habib F, Schulman CI, Duncan R, Proctor KG. Can near-infrared spectroscopy identify the severity of shock in trauma patients? J Trauma. 2005 Apr;58(4):806-13; discussion 813-6. doi: 10.1097/01.ta.0000158269.68409.1c. PMID 15824660
- [Background] Creteur J, Carollo T, Soldati G, Buchele G, De Backer D, Vincent JL. The prognostic value of muscle StO2 in septic patients. Intensive Care Med. 2007 Sep;33(9):1549-56. doi: 10.1007/s00134-007-0739-3. Epub 2007 Jun 16. PMID 17572876